CLINICAL TRIAL: NCT00907829
Title: Source of Neurally-Mediated Hand Weakness After Stroke
Brief Title: Source of Hand Weakness After Stroke
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Methods unexpectedly required additional refinement that precluded subject enrollment.
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B6302-W
Record Dates: First submitted 2009-05-21; First posted 2009-05-25 (Estimated); Last update posted 2014-05-05 (Estimated); Status verified 2014-05

CONDITIONS: Stroke; Cerebrovascular Accident
Keywords: stroke; fingertip force; muscle coordination
MeSH Terms: conditions — Stroke | interventions — Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Active Comparator): persons with severe hand impairment following hemiparetic stroke
  Interventions: Drug: lidocaine; Device: muscle stimulator
- Arm 2 (Active Comparator): persons with severe hand impairment following hemiparetic stroke
  Interventions: Device: muscle stimulator

INTERVENTIONS:
Drug: lidocaine — comparison of the effect of the drug to help improve finger function
  Arms: Arm 1
Device: muscle stimulator — comparison of the effect of stimulated muscle(s) on finger function

SUMMARY:
The purpose of this study is to determine whether neural block and neuromuscular electrical stimulation are effective in treating finger impairment due to stroke.

DETAILED DESCRIPTION:
The incidence of stroke-induced hemiparesis among veterans is likely to rise as this population ages. Post-stroke hemiparesis is often marked by persistent hand impairment, which adversely affects both a person's ability to work and his/her quality of life. We believe that impairment is primarily due to neural, rather than biomechanical, factors. At the muscle level, these factors relate either to the inability to activate muscles (i.e., low muscle activation) or to activate them appropriately (i.e., abnormal muscle co-activation). Currently it is unclear as to which one is largely responsible for weakness in the hand as the net mechanical effect, e.g., reduced fingertip force production, could be the same. Determination of voluntary muscle force generation could help to explain deficits in fingertip force production in specific directions, as well as to customize treatment approaches in which force generation ability of some muscles is decreased and others increased. The goal of this work is to explain the source of neurally-mediated weakness at the fingertip following hemiparetic stroke, and to design and experimentally test rehabilitation interventions that attempt to offset this weakness.

As we were refining the protocol to experimentally test a rehabilitation intervention-involving neural block and stimulation of select muscles to decrease and increase muscle force generation-it was more challenging than anticipated to locate, using ultrasound, small nerve branches to individual muscles for selective neural blocking. As a result we designed additional interventions, using a computer model, that reflected the physical limitation to implementation which could still hopefully lead to improved fingertip function. We are seeking novel approaches to locate and block small nerve branches to individual muscles for an individual muscle-based approach to rehabilitation which we expect to be an improvement over rehabilitation interventions that target groups of muscles at a time. The clinical data collected in the study and biomechanical model simulation work provide guidance for a clinical trial study in the future.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of stroke;
* stroke occurred no less than 6 months prior to study;
* must have had only 1 stroke;
* must demonstrate severe hand impairment;
* must have no substantial evidence of motor and sensory deficits in non-paretic limb;
* must have no history or clinical signs of neurologic diseases other than stroke;
* must have no cognitive dysfunction that precludes comprehension of experimental tasks;
* must be able to give informed consent

Exclusion Criteria:

* taking medication that can increase the risk of lidocaine toxicity such as cimetidine (ulcer treatment drug), phenytoin (anticonvulsant drug), nadolol (drug for treatment of headache, hypertension, chest pain);
* taking anticoagulant medication, i.e., aspirin, coumadin;
* has a low platelet count or a bleeding disease

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-02; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
fingertip force | force measured before and after intervention (1 week later)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Towles, Principal Investigator — Edward Hines Jr. VA Hospital
Locations (1):
- Edward Hines, Jr. VA Hospital, Hines, Illinois, United States